CLINICAL TRIAL: NCT00003391
Title: Phase I Trial of Monoclonal Antibody muJ591 in Patients With Hormone-Independent Prostate Cancer
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Prostate Cancer That Has Not Responded to Hormone Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Purpose: Treatment
Other Study IDs: CDR0000066389; NYH-CMC-0498-213; NCI-V98-1426
Record Dates: First submitted 1999-11-01; First posted 2004-07-22 (Estimated); Last update posted 2009-10-12 (Estimated); Status verified 2009-10

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Biological: monoclonal antibody muJ591

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of muJ591 monoclonal antibody in treating patients who have metastatic prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Define the toxicity and maximum tolerated dose of monoclonal antibody muJ591 in patients with hormone independent prostate cancer. II. Define the pharmacokinetics and biodistribution of monoclonal antibody muJ591 in these patients. III. Define the human antimouse antibody response to this therapy. IV. Define the preliminary efficacy of this therapy in these patients.

OUTLINE: This is a dose escalation study. Patients receive a single dose of intravenous iodine I 131-labeled monoclonal antibody muJ591 on day 0, combined with an unlabeled (cold) dose of monoclonal antibody muJ591. Anterior and posterior imaging is obtained 1 hour after labeled muJ591 administration and on days 0, 2, 4, and 6. Subsequent cohorts of 3-6 patients receive fixed iodine-labeled doses with escalating cold doses of monoclonal antibody muJ591 until the maximum tolerated dose is reached. Patients are followed for a minimum of 8 weeks after muJ591 therapy or until disease progression. Patients with stable or responding disease who are human anti-mouse antibody negative may receive subsequent treatments at the discretion of the principal investigator.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic adenocarcinoma of the prostate, defined by: Abnormal CT, MRI, or bone scan and/or Rising prostate specific antigen (PSA) levels (on 3 consecutive occasions over at least 6 weeks) despite hormonal therapy PSA at least 2.0 at study entry No active CNS metastases

PATIENT CHARACTERISTICS: Age: 21 and over Performance status: Karnofsky 60-100% Life expectancy: At least 6 months Hematopoietic: WBC greater than 3,500/mm3 Platelet count greater than 100,000/mm3 No serious hematologic disease Hepatic: SGOT less than 2.0 times upper limit of normal Bilirubin less than 1.5 mg/dL No serious hepatic disease Renal: Creatinine less than 2.0 mg/dL Calcium less than 13.5 mg/dL No serious renal disease Cardiovascular: No active angina No New York Heart Association class III-IV No other serious cardiac disease Pulmonary: No serious respiratory disease Other: No active uncontrolled infection Evidence of pre-existing antimouse antibody at the time of screening

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 6 weeks since prior cytotoxic chemotherapy Endocrine therapy: At least 6 weeks since prior adrenal hormone inhibitors or corticosteroid therapy Antiandrogen therapy must be discontinued prior to measuring PSA values Luteinizing hormone-releasing hormone analog must be maintained during study OR must be discontinued at least 10 weeks prior to study entry (for 28 day depot preparation) or 24 weeks prior to study entry (for 3 month depot preparation) Radiotherapy: At least 6 weeks since prior radiotherapy Surgery: Not specified

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1998-06

CONTACTS AND LOCATIONS:
Overall Officials: Neil H. Bander, MD, Study Chair — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital - Cornell Campus, New York, New York, United States

REFERENCES:
- [Derived] Vlachostergios PJ, Niaz MJ, Skafida M, Mosallaie SA, Thomas C, Christos PJ, Osborne JR, Molina AM, Nanus DM, Bander NH, Tagawa ST. Imaging expression of prostate-specific membrane antigen and response to PSMA-targeted beta-emitting radionuclide therapies in metastatic castration-resistant prostate cancer. Prostate. 2021 Apr;81(5):279-285. doi: 10.1002/pros.24104. Epub 2021 Jan 19. PMID 33465252